CLINICAL TRIAL: NCT06929975
Title: The Effect of Podcast Training on Birth Fear in Couples: A Randomized Controlled Trial
Brief Title: The Effect of Podcast Training on Birth Fear in Couples
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Betul Uncu, Lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/160
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Pregnancy; Birth Fear
Keywords: birth fear; pregnancy; podcast

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- podcast (Experimental): In accordance with the established training program for participants, a four-phase podcast listening process aimed at reducing birth fear will be implemented. The first podcast will be launched at the 33rd week of pregnancy, with the goal of helping participants gain information about the childbirth process and reduce their anxiety. Following that, a second podcast will be played at the 34th week of pregnancy, focusing on supporting psychological preparation for childbirth. The third podcast, to be implemented at the 35th week, will address topics such as relaxation techniques and breathing exercises that can be used during labor. Finally, the fourth podcast, played at the 36th week, will emphasize the importance of positive thinking and partner support during labor. To evaluate the effectiveness of the podcast sessions, psychological status and partner support scales will be applied at specific weeks.
  Interventions: Behavioral: podcast training
- control (No Intervention): Participants in the control group will not be provided with any podcast sessions; they will continue to benefit only from routine pregnancy follow-ups and existing healthcare services. This group will progress through the natural course without any special interventions, and standard prenatal care procedures will be applied. To measure changes in participants' birth fear and psychological conditions, data will be collected by applying specific scales at the 32nd, 37th, and 39th weeks of pregnancy. Additionally, the same scales will be used on the 2nd postpartum day to assess participants' psychological conditions after childbirth.

INTERVENTIONS:
Behavioral: podcast training — In accordance with the established training program for participants, a four-phase podcast listening process aimed at reducing birth fear will be implemented. The first podcast will be launched at the 33rd week of pregnancy, with the goal of helping participants gain information about the childbirth process and reduce their anxiety. Following that, a second podcast will be played at the 34th week of pregnancy, focusing on supporting psychological preparation for childbirth. The third podcast, to be implemented at the 35th week, will address topics such as relaxation techniques and breathing exercises that can be used during labor. Finally, the fourth podcast, played at the 36th week, will emphasize the importance of positive thinking and partner support during labor. To evaluate the effectiveness of the podcast sessions, psychological status and partner support scales will be applied at specific weeks.
  Arms: podcast

SUMMARY:
Birth fear refers to intense feelings of anxiety, fear, and worry regarding the childbirth process, often arising from concerns about physical pain, complications, or uncertainty about the baby's health. Many women experience this fear during pregnancy, which, in some cases, may develop into a clinical condition known as tokophobia . Birth fear can increase stress levels, disrupting the mother's hormonal balance, which may prolong labor, increase the risk of complications, and negatively impact fetal development. Additionally, it can lead to issues such as loss of self-confidence, anxiety, and depression in the mother, while causing communication problems and lack of support between partners. Birth fear affects not only the labor process but also the postpartum period, potentially leading to postpartum depression, trauma, and difficulties in mother-infant bonding. All these factors can adversely impact the psychosocial well-being of both women and couples. Therefore, it is crucial to develop interventions aimed at recognizing and reducing birth fear.

DETAILED DESCRIPTION:
Podcasts, with their accessibility, low cost, and user-friendly structure, allow individuals to access health-related information more easily and personalize the educational process, making it more effective. These factors make podcasts a valuable tool, especially in areas that require emotional and cognitive intervention, such as birth fear. While birth fear is a significant psychological factor influencing the anxiety of women and their partners regarding the childbirth process, there are limited intervention-focused studies targeting couples in this area. Although various methods have been proposed in the literature to reduce birth fear, data on the effectiveness of digital educational tools like podcasts in this domain is insufficient. This research aims to fill an important gap by evaluating the effect of a podcast series on birth fear in couples. The purpose of this study is to examine how a podcast series focused on birth fear impacts birth fear, anxiety, and postpartum depression in couples.

ELIGIBILITY:
Inclusion Criteria:

19-35 years old married primiparous 2nd trimester pregnant women

Exclusion Criteria:

Pregnant women with risky pregnancies illiteracy problems with internet access visual and hearing impairment

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 50 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-12-07 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Wijma Delivery Expectancy Questionnaire (W-DEQ) | 8 month
  This scale measures fear and expectations related to childbirth. Form A focuses on measuring fear of childbirth during pregnancy, while Form B assesses the postpartum process. The W-DEQ-A Form consists of 33 items. Low fear and anxiety are scored between 33-55 points, moderate fear and anxiety between 56-80 points, and high fear and anxiety between 81-165 points. It has three subscales: "Fear and Anxiety of Childbirth," "Expectations Regarding Childbirth," and "Emotional Responses to the Birth Process."
  The W-DEQ-B Form consists of 14 items across three subscales: "Fear of Childbirth," "Physical Reactions," and "Psychological Reactions." Low fear is scored between 14-28 points, moderate fear between 29-49 points, and high fear between 50-70 points.

SECONDARY OUTCOMES:
Tilburg Pregnancy Distress Scale: | 8 month
  This scale is used to determine the psychological stress and anxiety levels experienced during pregnancy. It measures individuals' negative feelings and thoughts regarding the pregnancy process. The scale is assessed through three subscales: "Emotional Distress," "Physical Distress," and "Social Support and Relationships." The total score reflects the intensity of the psychological and physical distress experienced by the individual during pregnancy. The total score determines the personal stress level. A score between 25-40 indicates low stress, between 41-60 indicates moderate stress, and a score of 61 and above indicates high stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Ağrı Training and Research Hospital, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data will not be shared due to privacy concerns and the protection of participant confidentiality. Additionally, there are no plans to make the data publicly available as the study is ongoing and the analysis is still in progress.

REFERENCES:
- [Background] Cai F, McCabe M, Srinivas SK. A randomized trial assessing the impact of educational podcasts on personal control and satisfaction during childbirth. Am J Obstet Gynecol. 2023 May;228(5):592.e1-592.e10. doi: 10.1016/j.ajog.2023.01.021. Epub 2023 Feb 13. PMID 36791987